CLINICAL TRIAL: NCT01806935
Title: Xerotic Dermatitis in Aged People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Medical Devices (Industry)
Responsible Party: Sponsor
Organization: Pierre Fabre Medicament (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-A01547-36
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-02

CONDITIONS: Itching Symptoms; Xerotic Dermatitis
Keywords: associated; aged population

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DC086 (Experimental): cream
  Interventions: Device: DC086
- placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: DC086
  Arms: DC086
Device: Placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to assess the the effect of the study product on itching symptoms associated with xerotic dermatitis in aged population

ELIGIBILITY:
Inclusion Criteria:

* Aged from 70 years
* With xerotic dermatitis, clinically assessed ,
* At least on the anterior part of lower and/or upper limbs,
* Presenting itching xerotic dermatitis evolving from at least 3 weeks
* Intensity of itching ≥ 4 on VAS (0-10) at th inclusion time
* With MMSE score ≥ 20 dating less than 6 months
* Affiliated to a social security system, or is a beneficiary (as applicable in the national regulation)

Exclusion Criteria:

* Criteria related to pathologies

  * Severe form of other dermatitis requiring either systemic treatment

    -- Itching xerotic dermatitis from iatrogenic origins
  * Dermatological disease other than xerotic dermatitis which could interfere with the assessment,
  * Systemic disease that may generate xerotic dermatitis and /or pruritus
  * Immunosuppression condition,
  * History of serious disease considered by the investigator hazardous for the patient or incompatible with the study.
* Criteria related to treatment

  - Use of treatment which could interfere with the evaluation of the disease or the course of the disease
* Criteria related to the population

  * Ongoing participation to another clinical trial or participation in the previous month before the inclusion
  * Patient under guardianship or trusteeship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Itching symptoms intensity change | From Day 1 to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yves Rolland, Principal Investigator — Hôpital Purpan CHU TOULOUSE, France
Locations (14):
- France (14):
  - 0521, Angers
  - 0523, Angers
  - 0520, Cugnaux
  - 0517, Le Fousseret
  - 0518, Muret
  - 0519, Muret
  - 0515, Saint-Orens-de-Gameville
  - 0516, Saint-Orens-de-Gameville
  - 0511, Seysses
  - 0512, Seysses
  - 0513, Seysses
  - 0514, Seysses
  - 0522, Tiercé
  - 0501, Toulouse